CLINICAL TRIAL: NCT05874453
Title: Effect of Evidence-Based Eye Care Protocol in Intensive Care Units
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Özlem Ceyhan, Assoc.Prof, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EYEPROTOCHOL
Record Dates: First submitted 2023-05-10; First posted 2023-05-25 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-02

CONDITIONS: Ocular Complications; Eye Protocol
Keywords: eye protocol; ocular complications; intensive care; nursing care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Eye care protocol to be appliedevaluation.
  Interventions: Other: eye care protocol
- Control Group (No Intervention): Routine intensive care Eye care protocol to be applied

INTERVENTIONS:
Other: eye care protocol — The lower conjunctiva of the eye to be treated is opened, 1-2 drops of gel are applied, the eye is closed. Cleaning eye secretions is done with sterile distilled water. A gel containing trehalose, hyaluronic acid and carbomer will be applied every 2-4 hours in accordance with intensive care eye care protocol. In order to determine the exposure keratopathy, staining with Fluorescein Sodium will be performed by the ophthalmologist on days 0, 5 and 10, and a blue light pen will be used for evaluation. In order to determine the degree of dry eye, the Schirmer I test will be performed on the 0th and 10th days
  Arms: Intervention Group

SUMMARY:
In intensive care patients, normal eye protection mechanisms such as tear production, blinking and keeping the eyes closed are impaired.

If eye-related complications are not diagnosed and treated in time, they can cause microbial keratitis and vision loss. This study was planned as a randomized controlled experimental study to examine the effect of using an evidence-based protocol on eye care on ophthalmologic complications. Patients who meet the inclusion criteria will be randomized, and one eye of the patients will be assigned to the intervention group (experimental group) and the other to the control group. When the study reaches 40 patients, G*Power analysis will be applied and the sample size will be decided according to the result.

ELIGIBILITY:
Inclusion Criteria:

* Patients connected to mechanical ventilator,
* Newly intubated patients,
* Patients who have not been diagnosed with keratopathy and keratoconjunctivitis as of hospitalization,
* Patients who have not been diagnosed with burns and facial injuries,
* Patients without chronic lagophthalmos and eye trauma before ICU admission

Exclusion Criteria:

* Patients who have received topical drug therapy other than ocular lubrication
* Patients with muscle weakness as a result of cranial nerve VII (facial) nerve palsy
* Patients with chronic lagophthalmos and eye infections
* Those with rheumatological diseases
* Those with neurological/neuropathic disease that will affect eye closure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Corneal Changes Rating Scale | the day before the intervention
  It is the diagnosis of ocular surface/corneal epithelial damage and dry eye syndrome by instillation of fluorescein sodium, which is used to determine corneal surface damage. A patient is considered to have exposure keratopathy if either eye has a grade greater than 0.
Corneal Changes Rating Scale | 5th day of application
  It is the diagnosis of ocular surface/corneal epithelial damage and dry eye syndrome by instillation of fluorescein sodium, which is used to determine corneal surface damage. A patient is considered to have exposure keratopathy if either eye has a grade greater than 0.
Corneal Changes Rating Scale | 10th day of application
  It is the diagnosis of ocular surface/corneal epithelial damage and dry eye syndrome by instillation of fluorescein sodium, which is used to determine corneal surface damage. A patient is considered to have exposure keratopathy if either eye has a grade greater than 0.

SECONDARY OUTCOMES:
Dry Eye Rating Scale | the day before the intervention
  The Schirmer I test is performed by placing the strip on the lower eyelid margin approximately 2 mm from the lateral canthus, away from the cornea. The eyelid is closed for five minutes and the wet portion of the strip is measured in millimeters. Values greater than 10 mm/5 minutes indicate the normal volume of the tear film
Dry Eye Rating Scale | 5th day of application
  The Schirmer I test is performed by placing the strip on the lower eyelid margin approximately 2 mm from the lateral canthus, away from the cornea. The eyelid is closed for five minutes and the wet portion of the strip is measured in millimeters. Values greater than 10 mm/5 minutes indicate the normal volume of the tear film
Dry Eye Rating Scale | 10th day of application
  The Schirmer I test is performed by placing the strip on the lower eyelid margin approximately 2 mm from the lateral canthus, away from the cornea. The eyelid is closed for five minutes and the wet portion of the strip is measured in millimeters. Values greater than 10 mm/5 minutes indicate the normal volume of the tear film

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Hospital, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Background] El Hachimi R, El Hadiri R, Benchekroun S, Boutimzine N, Amazouzi A, Cherkaoui LO, Maazouzi AW. [Incidence and risk factors of exposure keratopathy in intensive care units: About 91 patients]. J Fr Ophtalmol. 2022 Dec;45(10):1137-1143. doi: 10.1016/j.jfo.2022.03.009. Epub 2022 Oct 29. French. PMID 36319529
- [Background] Ezra DG, Chan MP, Solebo L, Malik AP, Crane E, Coombes A, Healy M. Randomised trial comparing ocular lubricants and polyacrylamide hydrogel dressings in the prevention of exposure keratopathy in the critically ill. Intensive Care Med. 2009 Mar;35(3):455-61. doi: 10.1007/s00134-008-1284-4. Epub 2008 Sep 23. PMID 18810388
- [Background] Hartford JB, Bian Y, Mathews PM, De Rojas J, Garg A, Rasool N, Schroder SK, Trief D. Prevalence and Risk Factors of Exposure Keratopathy Across Different Intensive Care Units. Cornea. 2019 Sep;38(9):1124-1130. doi: 10.1097/ICO.0000000000001961. PMID 31394552
- [Background] Kousha O, Kousha Z, Paddle J. Exposure keratopathy: Incidence, risk factors and impact of protocolised care on exposure keratopathy in critically ill adults. J Crit Care. 2018 Apr;44:413-418. doi: 10.1016/j.jcrc.2017.11.031. Epub 2017 Nov 28. PMID 29353117
- [Background] Mela EK, Drimtzias EG, Christofidou MK, Filos KS, Anastassiou ED, Gartaganis SP. Ocular surface bacterial colonisation in sedated intensive care unit patients. Anaesth Intensive Care. 2010 Jan;38(1):190-3. doi: 10.1177/0310057X1003800129. PMID 20191796